CLINICAL TRIAL: NCT03884985
Title: Eye Movements, Visual Perception and Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Martina Poletti, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RSRB00069578; R01EY029788-01 (NIH)
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Vision
MeSH Terms: interventions — Photic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal Vision (Experimental): This study examines high-acuity vision, oculomotor behavior recorded using high-resolution eyetracking. Healthy participants are asked to perform different types of visual tasks, ranging from letter identification to judging facial expressions while their eye movements will be recorded with high-precision together with their behavioral performance in the task.
  Interventions: Other: Visual stimulation

INTERVENTIONS:
Other: Visual stimulation — In the experiments, participants will sit in front of a computer monitor located a less than a meter of distance and will analyze the content of images extracted from collections of natural and computer-generated scenes. Subjects will be asked to report verbally or by pressing keys on a keyboard on image characteristics such as the locations of the objects present in the scenes, their number and/or their identities. Some experiments will involve a search paradigm in which subjects will have to report on the location and/or fine characteristics of a target element among a field of distracting similar elements, and/or visual discrimination tasks. The duration of the interval of time in which the image is maintained on the screen may be varied between few tens of milliseconds to several seconds. In a set of experiments, the eye movements performed by the subjects during the execution of the visual tasks will be recorded as explained below.

SUMMARY:
During visual fixation, small eye movements of which we are usually not aware, prevent the maintenance of a steady direction of gaze. These eye movements are finely controlled and shift retinal projection of objects within the fovea, the region of the retina where visual acuity is highest. This program of research examines the link between these eye movements and attention, and tests the hypothesis that attention, similarly to eye movements, can be controlled at the foveal level. Psychophysical experiments with human subjects, using state-of-the-art techniques, high resolution eyetracking and retinal stabilization are conducted to address these questions. Gaze-contingent calibration procedures are employed to achieve high accuracy in gaze localization. A custom developed gaze-contingent display is used to shift in real-time visual stimuli on the monitor to compensate for the observer eye movements during fixation periods and to maintain stimuli at a desired location on the retina. Experiments involve visual discrimination/detection tasks with stimuli presented at selected eccentricities within the fovea. Participants' performance and reaction times are examined under different conditions, in which various types of attention are manipulated. In addition to advancing our basic understanding of visual perception, this research leads to a better understanding of attentional control at the foveal scale and of the contribution of microscopic eye movements to the acquisition and processing of visual details.

DETAILED DESCRIPTION:
The goals of this study are to the following:

1. Examine the resolution and time-course of attention within the foveola. Attentional control has been traditionally studied outside the foveola but the PI's recent work suggests that attentional shifts also play a critical role in the normal examination of fine spatial details. Building on our previous results, we will investigate the extent by which both voluntary and involuntary attention can be controlled at this scale. Specifically, we will (a) measure the resolution of attention, i.e., the minimum distance between two locations within the foveola that can elicit selective voluntary attentional shifts. We will (b) examine whether enhancements in fine spatial vision at selected foveal locations, such as those we have previously shown for voluntary attention, also occur with involuntary attention. Finally we will study (c) the time-course of attentional enhancements and inhibition of return at this scale. Moreover, to study how peripheral and foveal attention differ, we will compare the extent of exogenous attentional effects and their time-course within and outside the foveola.
2. Map visual acuity and crowding across the foveola. Our research has shown that vision is not uniform across the foveola: discrimination of fine spatial patterns is already suboptimal just a few arcmins away from the center of gaze. This phenomenon could be caused by a decline in visual acuity outside the preferred retinal locus and/or the consequences of crowding, the negative influence resulting from objects adjacent to the target. Because of the difficulty in precisely controlling retinal stimulation at this scale, it is unclear whether crowding occurs in the foveola, and whether its influence changes with foveal eccentricity. We will measure both visual acuity (a), and crowding (b), and will assess their relative contribution over a range of foveal eccentricities, both nasally and temporally. In addition to examine visual acuity across subjects, we will also examine how it changes at the individual level.
3. Link attention, fine spatial vision and oculomotor control. Microsaccades normally shift the retinal projection of the fixated object across the foveola. At a larger scale, visual resolution, attention, and eye movements are tightly coupled. But little is known on whether and how this interplay unfolds within the foveola. Here we will investigate how attention and vision interact with microsaccades preparation and execution. We will examine (a) whether microsaccades preparation yields attentional benefits at specific foveal locations; (b) the precision of microsaccades; (c) their impact in attenuating negative effects of reduced acuity and foveal crowding, and; (d) their impact on performance in natural high acuity tasks.

To address these goals psychophysics experimental paradigms and high-precision eyetracking will be used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for the study if they:

  * Are at least 18 years old
  * Speak English
  * Have read, understood, and signed the informed consent form Have normal visual acuity (20/20 or better) without correction (i.e. without glasses or contact lenses) and no known visual deficits. A standard visual acuity screening will be performed by means of a Snellen chart (the standard eye chart) at the beginning and the end of the experiments.

Exclusion Criteria:

* Subjects will be excluded if they:

  * Are under 18 years old
  * Cannot understand the experimental procedures Have reported vision loss, including the need for correction (i.e. glasses or contact lenses), or fail the visual acuity screening performed during the experiments. We expect a very minor portion of subjects to be excluded as a result of this test, as the good vision requirement will be clearly stated in our recruitment materials. There will be no data collection for subjects who will not pass the acuity test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martina Poletti, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Vision
Started | 155
Completed | 155
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Normal Vision
Number analyzed (Participants) | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 155
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 43
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 73
  More than one race | 15
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 155

OUTCOME MEASURES:

1. Primary Outcome: Average Performance in Visual Tasks
Description: Proportion correct responses in visual tasks. For each visual stimulus presentation, observers performed a four-alternative forced-choice (4AFC) task. A trial was considered correct if the participant's selected response matched the identity of the presented stimulus; otherwise, it was marked as incorrect.
Time Frame: Day 0
Population: Percent correct responses in visual tasks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Normal Vision
Number analyzed (Participants) | 155
percentage | 74 (9)

2. Primary Outcome: Microsaccades Rate
Description: rate of microsaccades per second
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: microsaccades per second
Arm/Group | Normal Vision
Number analyzed (Participants) | 155
microsaccades per second | 0.5 (0.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected right after each experimental session. No adverse event occurred. This is a minimal risk study.
Arm/Group | Normal Vision
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT03884985/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT03884985/ICF_001.pdf